CLINICAL TRIAL: NCT01677468
Title: Phase Study About Feeding Artery Obliteration by Chemoembolization on Survival of Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Survival According to the Feeding Artery Obliteration by Chemoembolization for Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-12-122
Record Dates: First submitted 2012-08-09; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Hepatocellular Carcinoma; Transarterial Chemoembolization
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin; Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermediate embolization (Experimental): TACE with substatsis using gelfoam
  Interventions: Procedure: Intermediate embolization
- Complete embolization (Active Comparator): TACE with complete embolization using gelfoam
  Interventions: Procedure: Complete embolization

INTERVENTIONS:
Procedure: Intermediate embolization — TACE with substasis using gelfoam
  Other Names: Adriamycin; Cysplatin; Gelfoam
  Arms: Intermediate embolization
Procedure: Complete embolization — TACE with complete embolization using gelfoam
  Other Names: Adriamycin; Cysplatin; Gelfoam
  Arms: Complete embolization

SUMMARY:
The aim of this study was to evaluate whether survival of patients who underwent TACE with unresectable HCC can benefit from intermediate-levels of embolization.

DETAILED DESCRIPTION:
Subjective angiographic chemoembolization endpoints (SACE) levels were developed to standardize the embolic endpoints of transarterial chemoembolization (TACE) for hepatocellular carcinoma (HCC). It determined the antegrade arterial flow and residual tumor blush as follows: I, normal-normal; II, reduced-reduced; III, reduced-none; IV, none-none. SACE level II and III indicates intermediate-levels of embolization, whereas IV indicates overembolization. The aim of this study was to evaluate whether survival of patients who underwent TACE with unresectable HCC can benefit from intermediate-levels of embolization.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* ECOG performance status 0-2
* Hepatocellular carcinoma diagnosed histologically or clinically
* Tumor numbers of 5 or less
* No history of treatment for hepatocellular carcinoma
* Patients with informed consent

Exclusion Criteria:

* Extrahepatic metastasis
* Rupture of hepatocellular carcinoma
* Infiltrative hepatocellular carcinoma
* Malignancy other than hepatocellular carcinoma

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Survival rate of the subjects | 6 months after TACE
  Survival rate of the subjects 6 months after TACE
Survival rate of the subjects | 12 months after TACE
  Survival rate of the subjects, 12 months after TACE
Survival rate of the subjects | 18 months after TACE
  Survival rate of the subjects, 18 months after TACE
Survival rate of the subjects | 24 months after TACE
  Survival rate of the subjects, 24 months after TACE

SECONDARY OUTCOMES:
Disease free survival of the subjects | 6, 12, 18, and 24 months after TACE
  Disease free survival of the subjects, 24 months after TACE
Complication rate of TACE | 6, 12, 18, and 24 months after TACE
  The incidence of infection, hemorrhage, 24 months after TACE

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Park, M.D., Ph.D., Principal Investigator — Hallym University Medical Center
Locations (3):
- South Korea (3):
  - Hallym Sacred Heart Hospital, Anyang
  - Chuncheon Sacred Heart Hospital, Chuncheon
  - Kangnam Sacred Heart Hostpita, Seoul